CLINICAL TRIAL: NCT01617941
Title: A Multi-center, Randomized, Double-blind, Parallel Group, Placebo Controlled, Study in Patients With Non-chronic Migraine to Assess the Efficacy, Safety and Tolerability of BID Oral Doses of BGG492 in Migraine Prevention.
Brief Title: A Randomized,Double Blind, Placebo Controlled Study to Assess Efficacy,Safety and Tolerability of BGG492 in Migraine Prevention
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBGG492A2214; 2011-005316-28 (EudraCT Number)
Record Dates: First submitted 2012-06-10; First posted 2012-06-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-09

CONDITIONS: Patients With Migraine Equal of /More Than 3 and Equal of/ Less Than 12 Migraine Attacks/4 Weeks for Each of the Last 6 Months Preceding the Screening
Keywords: non-chronic migraine, migraine prevention
MeSH Terms: interventions — selurampanel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BGG492 (Experimental): At Baseline 60 patients will be randomized to receive BGG492 for the upcoming 12 weeks (dose: 75 mg BID administered in approx. 12 hours +/- 2 hours intervals).
  Interventions: Drug: BGG492
- Placebo (Placebo Comparator): At Baseline 30 patients will be randomized to receive Placebo for the upcoming 12 weeks (matching a dose of 75 mg BID BGG492 administered in approx. 12 hours +/- 2 hours intervals).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGG492
  Arms: BGG492
Drug: Placebo — In patients not tolerating a dose of 75 mg BID BGG492/Placebo the dose can be decreased to 50 mg BID and this dose will be continued for the rest of the planned treatment. Those patients who are not tolerating 50 mg BID BGG492/Placebo will be discontinued from the trial.
  Arms: Placebo

SUMMARY:
It will provide a first evaluation of efficacy, safety and tolerability of BGG492 in patients with non-chronic migraine having more than 3 and less than 12 migraine attacks per 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female smoking and non-smoking subjects of 18 to 65 years of age (inclusive)
* Patients diagnosed with non-chronic migraine with or without aura of duration of at least 12 months prior to the study start
* Patient diagnosed with migraine (according to the International Headache Society categories 1.1 and with equal to/more than 3 and equal to/ less than 12 migraine attacks per 4 weeks for each of the last 6 months preceding the Screening
* Patients willing to abstain from activities that require focused attention, e.g. driving a car or other vehicles, operating machines or engaging in potentially dangerous activities that require focused attention and intact physical balance

Exclusion Criteria:

* Patients diagnosed with basilar, ophthalmoplegic or hemiplegic migraine as shown in the current/past medical history.
* Patients having an experience of non-migraine headaches on more than 6 days per 4 weeks in the past 6 months prior to study start
* Patients receiving regular treatment during the four (4) weeks preceding the Baseline with psychoactive drugs (e.g. hypnotics, benzodiazepines, neuroleptics) except antidepressants (eg. SSRIs, SNRIs, Tri- or Tetracyclics).
* Patients receiving migraine prevention medications during past three (3) months preceding Baseline
* Patients receiving topiramate as migraine prevention medication during past six (6) months preceding Baseline
* Patients receiving metamizole as acute treatment of migraine during past three (3) months preceding Baseline
* Patients using (or having used within four (4) weeks before the treatment start) drug treatments that are potent inhibitors of OATP transporters (e.g. rifampin).
* Any psychiatric condition (e.g., schizophrenia, dementia, bipolar disorder) as shown in the past medical history prior to study start
* Patients with recent (within the last three [3] years prior to study start) and/or recurrent history of autonomic dysfunction (e.g. recurrent episodes of fainting, palpitations, orthostatic hypotension etc.).
* Pregnant or nursing (lactating) women. Baselines (1 and 2).
* Patients with history of drug or alcohol abuse within the 12 months prior to dosing Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of migraine attacks | 12 weeks
  50% responder rate (equal to or more than 50 % reduction in attack frequency during the last 4-weeks of the 12-weeks treatment period compared with the 4-weeks Baseline period)

SECONDARY OUTCOMES:
Number of migraine attacks | 12 weeks
  Mean change in number of migraine attacks comparing the last 4-weeks treatment with the Baseline period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals